CLINICAL TRIAL: NCT03225430
Title: Evaluation of a Cognitive Psychophysiological Treatment for Tourette Syndrome and Tic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Frederick Aardema, Professeur titulaire, Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 340559
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Tic Disorder, Chronic Motor or Vocal; Tourette Syndrome in Children; Tourette Syndrome
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors will receive no information on participant history and psychopathology. All evaluation sessions will be audio-recorded for reliability and to ensure that treatment status is not divulged. The Assessors will be separated from the therapists by geographical location site and will sign agreements not to discuss cases in the study with any other team member. Child and adult participants will agree not to discuss treatment or therapy during evaluation. Management of assessors will be delegated to a separate clinical coordinator who will assume overall responsibility for evaluations and preempting any direct contact between the principal investigator and Co-investigators and the assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Behavioural Intervention (Active Comparator): Participant will received psychoeducation about tic disorders, creating a tic hierarchy that will be revised during future sessions, introduce concept of function-based intervention, behavioral reward program, self-monitoring training, habit reversal training for their tics. They will received an introduction of relaxation techniques and diaphragmatic breathing exercise and an introduction of progressive muscle relaxation (PMR) exercise.
  They will received booster sessions for three months and he will do hierarchy review, inconvenience review, function-based intervention and competing response review, review of relaxation techniques and relapse prevention review.
  Interventions: Behavioral: Cognitive behavioural treatment for tics
- Cognitive psychophysiological (CoPs) (Experimental): The participant will received a rational about the treatment and awareness training about tics and creating list of tics. He will identifying high and low risk situations provoking tics, do video record and make a list of inconveniences of tic. He will do a screening session of the video and muscle discrimination exercises. Worked on a situational profile with a Kelly's grill and beginning relaxation and breathing exercises. He will identifying style of planning and work on it to do an advantages and inconveniences list to adopt this style. Some behavioral and cognitive re structuration about style of planning and how to modifying. At the end, he will received a relapse prevention informations and how to generalize the learnings and a record of the therapy. Finally, he will have to practice all this techniques at home for four week and do a last session to discuss home practice and received strategies for the future.
  Interventions: Behavioral: Cognitive psychophysiological

INTERVENTIONS:
Behavioral: Cognitive behavioural treatment for tics — Mainly based on the habit reversal treatment (HRT) and in addition to HRT components, they learn awareness training, relaxation, competing response, contingency management, and generalization training.
  Other Names: CBIT
  Arms: Comprehensive Behavioural Intervention
Behavioral: Cognitive psychophysiological — Focus on the processes influencing thoughts and behaviors underlying tics.
  Other Names: CoPs
  Arms: Cognitive psychophysiological (CoPs)

SUMMARY:
It is a randomized controlled trial to compare two behavioural treatments, namely CBIT and CoPs. This study would be the first head-to-head randomized trial between two established treatments rather than supportive counseling or wait-list control. Thirty-six adults and 36 children with TS/TD will be recruited into each of the two (CBIT, CoPs) modalities requiring a total recruitment of 72 adults and 72 children over 5 years, which permits, even for a small-medium effect size, a robust power calculation. Motor performance measures will give concurrent validity to changes pre-post in TS/TD motor processes. Recruitment of both males and females will permit sex comparisons. The participants meeting inclusion/exclusion criteria will be assessed at pre-post 1 month and 6 months following treatment on standardized tic scales and global assessment of functioning. Participants will be treated individually on a weekly basis by therapists with an allegiance to each modality and outcome assessed by masked evaluation. The treatments are manualized and will last 10 weeks with 4 weeks of home practice at post-treatment with 6-month follow-up assessment on all outcome measures, plus motor performance measures post-treatment. All treatment sessions will be audio-recorded and assessed with implementation of treatment integrity procedures scales. The hypotheses are that: (1) the CoPs group will show superiority in clinically significant improvement on standard tic scale score, global functioning and quality of life than the CBIT group; and (2) changes in recognized parameters on selected motor tests scored according to published norms will change towards normalization post CoPs but not post CBIT. The outcome data from the two treatments will be analyzed by a mixed linear model adaptation of repeated measures MANOVA and daily diary measures will allow for an additive time series design over the 10 weeks treatment session. This design will allow computation of the size of treatment effects at different stages of therapy. The study results will impact on the treatment of choice and access to treatment for tic disorders and on the conceptualization of tic disorders.

DETAILED DESCRIPTION:
Tics are defined as repetitive non-voluntary contractions of functionally related groups of skeletal muscles in one or more parts of the body. Gilles de la Tourette's syndrome (TS) forms a separate diagnostic category with multiple tics including vocal (phonic) tics occurring several times per day, for at least 1 year with onset before age 18. Persistent (chronic) tic disorder (TD) may involve a single motor or vocal tic. Tics peak around age 11 but can persist into adulthood with a prevalence of 1% and if untreated cause significant impairment. The current treatment guidelines for managing the tics recommend a Behavioural treatment, "habit reversal", which focuses on reversing the tic habit, now developed as a Comprehensive Behavioural Intervention for Tics (CBIT). CBIT involves multiple stages including awareness, relaxation, contingency training, positive reinforcement for not do the tic and the practice of a competing response antagonistic to the tic. A recent large scale multisite study compared CBIT with supportive therapy and found a significantly greater decrease in adults and children tics treated with CBIT. However, in both adult and child studies, 48-62% of samples were classified as non-responders. Effect sizes were medium (Cohen's d´= 0.55 - 0.68) compared to supportive therapy with mean tic decrease of 25-30% and samples remained symptomatic at follow-up. Research over the last 10 years (funded by the CIHR) have led to elaboration of a cognitive behavioural psychophysiological model of treatment (CoPs) of tic disorders. The CoPs is multi-modal and targets cognitive, behavioural and physiological processes characteristic of tic disorders rather than focusing on reversing the actual tic at onset. In the last funding period 2009-2013 the investigators have successfully applied the program to all subtypes and severity of adults with TS/TD both with and without comorbidity and compared outcome with a natural waitlist control. Results showed a clinically significant reduction of tic frequency following CoPs (Cohen's d- 1.43-2.34), maintained at 6-month follow-up. Validity of the CoPs model was supported by a change in behavioural and psychosocial as well as tic symptom measures post-treatment and at 6-month follow-up, and a post-treatment normalization of participants' performance on neuropsychological and electrophysiological measures.

ELIGIBILITY:
Inclusion Criteria:

* presenting a simple/complex tic for at least one year occurring daily. Those included in the TS group, age 8-12 or 18-65, had a diagnosis of TS as the principal presenting problem accompanied by vocal tics. Those included in the TD group presented a simple/complex tic (vocal or motor) for at least one year occurring daily.

Exclusion Criteria:

* any major medical history, head injury including sensori-motor impairment, history of autism, Intelligence Quotient (IQ)<75; other psychiatric problem on Axis I or II requiring treatment (minor comorbidities were accepted), any neurological problems (e.g., Parkinson's, hemifacial spasms, Meige syndrome, sclerosis; Huntington's disease, Wilson's disease); currently receiving treatment from a psychologist, acupuncture, hypnotherapist, massotherapist; currently receiving psychotropic drugs non-relevant to TS or ADHD or abuse of alcohol or drugs.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-04-21 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | baseline
  The YGTSS is a clinician-rated scale used to assess change in tic severity and impairment due to tics.

SECONDARY OUTCOMES:
determine style of planning actions | baseline
  The style of planning (STOP) questionnaire was developed to assess everyday style of planning actions. The aim of the STOP was to capture the behavioural and cognitive aspects involved in adequate planning of action in a variety of everyday situations involving routing, complex tasks and both anticipation and enactment.
measure effect of therapy in style of planning score | change from baseline
  The style of planning (STOP) questionnaire was developed to assess everyday style of planning actions. The aim of the STOP was to capture the behavioural and cognitive aspects involved in adequate planning of action in a variety of everyday situations involving routing, complex tasks and both anticipation and enactment.
measure long term effect of therapy in style of planning score | change from baseline at 6 months
  The style of planning (STOP) questionnaire was developed to assess everyday style of planning actions. The aim of the STOP was to capture the behavioural and cognitive aspects involved in adequate planning of action in a variety of everyday situations involving routing, complex tasks and both anticipation and enactment.
change in dimensions of perfectionism and use as a predictive variable of treatment issues | baseline
  The Frost Multidimensional Perfectionism Scale is a self-administered questionnaire of 35 items covering six dimensions of perfectionism.
change in dimensions of perfectionism | change from baseline
  The Frost Multidimensional Perfectionism Scale is a self-administered questionnaire of 35 items covering six dimensions of perfectionism.
measure the long term effect on dimensions of perfectionism | change from baseline at 6 months
  The Frost Multidimensional Perfectionism Scale is a self-administered questionnaire of 35 items covering six dimensions of perfectionism.
determine the initial score of symptom of anxiety use as a predictive variable of treatment issues | baseline
  The Beck Anxiety Inventory consists of a 21-item anxiety symptom checklist rating symptom intensity for the last week on a 0-3 scale.
measure the effect of therapy on symptom of anxiety | change from baseline
  The Beck Anxiety Inventory consists of a 21-item anxiety symptom checklist rating symptom intensity for the last week on a 0-3 scale.
measure the long term effect of therapy on symptom of anxiety | change from baseline at 6 months
  The Beck Anxiety Inventory consists of a 21-item anxiety symptom checklist rating symptom intensity for the last week on a 0-3 scale.
determine an initial score of symptom of depression and use as a predictive variable of treatment issues | baseline
  The Beck Depression Inventory consists of a 21-item relative to depression (α = .91), assesses cognitive, emotional and somatic depressive symptoms.
measure the effect of therapy on symptom of depression | change from baseline
  The Beck Depression Inventory consists of a 21-item relative to depression (α = .91), assesses cognitive, emotional and somatic depressive symptoms.
measure the long term effect of therapy on symptom of depression | change from baseline at 6 months
  The Beck Depression Inventory consists of a 21-item relative to depression (α = .91), assesses cognitive, emotional and somatic depressive symptoms.
measure the presence and the impact on treatment issues of major life events | baseline
  Life Events Survey determine which life events have occurred in the participant life over the past two years.
measure the presence and the impact on treatment issues of major life events | change from baseline
  Life Events Survey determine which life events have occurred in the participant life over the past two years.
measure the presence and the impact of major life events | change from baseline at 6 months
  Life Events Survey determine which life events have occurred in the participant life over the past two years.
determine an initial score of individual self-esteem and use as a predictive variable of treatment issues | baseline
  The Self-Esteem Inventory measure individual self-esteem
measure the effect of the therapy on Self-Esteem | change from baseline
  The Self-Esteem Inventory measure individual self-esteem
measure the long term effect of the therapy on Self-Esteem and use as a predictor of issues of treatment | change from baseline at 6 months
  The Self-Esteem Inventory measure individual self-esteem
determine an initial score of individual motor and attentional impulsivity and use as a predictive variable of treatment issues | baseline
  Barrat Impulsivity Scale measure motor and attentional impulsivity
measure the effect of the therapy on motor and attentional impulsivity | change from baseline
  Barrat Impulsivity Scale measure motor and attentional impulsivity.
measure the long term effect of the therapy on motor and attentional impulsivity | change from baseline at 6 months
  Barrat Impulsivity Scale measure motor and attentional impulsivity.
determine a baseline score of quality of life linked with Tourette syndrome | baseline
  Tourette syndrome quality of life questionnaire measure change in quality of life linked with symptoms of Tourette syndrome
measuring effect of therapy on quality of life | change from baseline
  measure change in quality of life linked with symptoms of Tourette syndrome
measuring long term effect of therapy on quality of life | change from baseline at 6 months
  measure change in quality of life linked with symptoms of Tourette syndrome
measuring initial symptoms of ADHD and use as a predictive variable of treatment issues | baseline
  The Conners Adult and child ADHD Rating Scale - Short: Self-administered is a self-reported questionnaire which measures attention deficit hyperactivity disorder (ADHD) symptoms.
measuring effect of therapy on symptoms of ADHD | change from baseline
  The Conners Adult ADHD Rating Scale - Short: Self-administered is a self-reported questionnaire which measures ADHD symptoms.
measuring long term effect of therapy on symptoms of ADHD | change from baseline at 6 months
  The Conners Adult ADHD Rating Scale - Short: Self-administered is a self-reported questionnaire which measures ADHD symptoms.
assessing symptom severity of obsessive-compulsive disorder (OCD) and use as a predictive variable of treatment issues | baseline
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) is assessing symptom severity in older children (i.e., 8-18 years) diagnosed with obsessive-compulsive disorder (OCD).
assessing change of symptom severity of obsessive-compulsive disorder (OCD) | change from baseline
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) is assessing symptom severity in older children (i.e., 8-18 years) diagnosed with obsessive-compulsive disorder (OCD).
assessing long term change of symptom severity of obsessive-compulsive disorder (OCD) | change from baseline at 6 months
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) is assessing symptom severity in older children (i.e., 8-18 years) diagnosed with obsessive-compulsive disorder (OCD).
determine an initial score of level of self-esteem use as a predictive variable of treatment issues | baseline
  The Culture Free Self-Esteem inventory is a self-report inventories used to determine the level of self-esteem in students ages 6-18 years and adults. It can be used to identify children and adolescents or adults in need of psychological assistance due to self-esteem problems, assess therapeutic progress, and evaluate post-therapy effects.
evaluate post-therapy effects on level of self-esteem | change from baseline
  The Culture Free Self-Esteem inventory is a self-report inventories used to determine the level of self-esteem in students ages 6-18 years and adults. It can be used to identify children and adolescents or adults in need of psychological assistance due to self-esteem problems, assess therapeutic progress, and evaluate post-therapy effects.
evaluate long term post-therapy effects on level of self-esteem | change from baseline at 6 months
  The Culture Free Self-Esteem inventory is a self-report inventories used to determine the level of self-esteem in students ages 6-18 years and adults. It can be used to identify children and adolescents or adults in need of psychological assistance due to self-esteem problems, assess therapeutic progress, and evaluate post-therapy effects.
change in the global measure of level of functionning in children, adolescents and adults | baseline
  The Childrens Global Assessment Scale (CGAS) and the global assessment scale (GAS) they are global measures of level of functioning in children and adolescents and adult. This measures provides a single global rating only, on scale of 0-100. In making their rating, the clinician makes use of the glossary details to determine the meaning of the points on the scale.
change in the global measure of level of functionning in children, adolescents and adults | change from baseline
  The Childrens Global Assessment Scale (CGAS) and the global assessment scale (GAS) they are global measures of level of functioning in children and adolescents and adult. This measures provides a single global rating only, on scale of 0-100. In making their rating, the clinician makes use of the glossary details to determine the meaning of the points on the scale.
change in the global measure of level of functionning in children, adolescents and adults | change from baseline at 6 months
  The Childrens Global Assessment Scale (CGAS) and the clinical global assessment of functionning scale (GAF) are global measures of level of functioning in children and adolescents and adult. This measures provides a single global rating only, on scale of 0-100. In making their rating, the clinician makes use of the glossary details to determine the meaning of the points on the scale.

OTHER OUTCOMES:
Intelligence and executive functioning screening assessment | baseline
  General intelligence evaluation with subscales of the Wechsler Adult Intelligence Scale or the Wechsler Intelligence Scale for Children, (WAIS-III or WISC-V - Vocabulary, block and similitude).
Intelligence and executive functioning screening assessment | change from baseline
  General intelligence evaluation with subscales of the Wechsler Adult Intelligence Scale or the Wechsler Intelligence Scale for Children, (WAIS-III or WISC-V - Vocabulary, block and similitude).
The Brief Inventory of Executive Function (BRIEF-A) | baseline
  Is a standardized 75-item questionnaire designed to assess adult's and children's views of their everyday environment.
The Brief Inventory of Executive Function (BRIEF-A) | change from baseline
  Is a standardized 75-item questionnaire designed to assess adult's and children's views of their everyday environment.
Motor function | baseline
  The assessment of fine motor dexterity by the Purdue pegboard test and for the evaluation of motor speed and control, the finger tapping task will be administered.
Motor function | change from baseline
  The assessment of fine motor dexterity by the Purdue pegboard test and for the evaluation of motor speed and control, the finger tapping task will be administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche de l'Institut universitaire en santé mentale de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No